CLINICAL TRIAL: NCT05167162
Title: Efficacy of the Most Commonly Used Physiotherapeutic Treatments for Acute Lower Limb Fatigue in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Gema Leon (Other)
Responsible Party: Principal Investigator, GEMA LEÓN BRAVO, Principal Investigator, Clinica Gema Leon
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ART-GLB-ACUTE FATIGUE
Record Dates: First submitted 2021-11-06; First posted 2021-12-22 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Lower Limb Injury
Keywords: Lower limbs; Physiotherapy; Athlete; Biomechanics; Protocol
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Intervention Model Description: 80 patients divided into 4 groups of equal size and randomly selected. The 4 treatment methods used will be as follows:
  Group 1: Compression techniques (n=20). Group 2: Massage techniques (n=20) Group 3: Hydrotherapy (n=20) Group 4: Active recovery technique (n=20)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Compression technique (Active Comparator): 20 participants make up the compression technique group.
  Interventions: Diagnostic Test: State-Trait Anxiety Questionnaire; Diagnostic Test: Rating of Perceived Exertion; Diagnostic Test: Motor coordination tests; Procedure: Physiotherapeutic intervention; Other: Data Analysis
- Group 2: Massage techniques (Active Comparator): 20 participants make up the massage technique group.
  Interventions: Diagnostic Test: State-Trait Anxiety Questionnaire; Diagnostic Test: Rating of Perceived Exertion; Diagnostic Test: Motor coordination tests; Procedure: Physiotherapeutic intervention; Other: Data Analysis
- Group 3: Hydromassage (Active Comparator): 20 participants make up the hydromassage technique group.
  Interventions: Diagnostic Test: State-Trait Anxiety Questionnaire; Diagnostic Test: Rating of Perceived Exertion; Diagnostic Test: Motor coordination tests; Procedure: Physiotherapeutic intervention; Other: Data Analysis
- Group 4: Active recovery technique. (Active Comparator): 20 participants make up the active recovery technique group.
  Interventions: Diagnostic Test: State-Trait Anxiety Questionnaire; Diagnostic Test: Rating of Perceived Exertion; Diagnostic Test: Motor coordination tests; Procedure: Physiotherapeutic intervention; Other: Data Analysis

INTERVENTIONS:
Diagnostic Test: State-Trait Anxiety Questionnaire — The scale measures ordinally (1 to 5) the values observed during exposure to anxiety patterns during exercise, such as higher repetitions, greater weight gain or longer exercise duration, as follows:
  1. Not at all
  2. Little
  3. Sometimes
  4. Almost always
  5. Always
  Other Names: STAI
Diagnostic Test: Rating of Perceived Exertion — The scale measures in ordinal form (1 to 6) the perceived effort during the exercise as follows:
  1. No pain
  2. Little pain
  3. Moderate
  4. Severe
  5. Very strong
  6. Unbearable
  Other Names: RPE
Diagnostic Test: Motor coordination tests — The motor coordination tests are divided into three:
  1. Jumping with 2 feet together.
  2. Throwing 2 balls from a given distance and space.
  3. Proprioception turns
Procedure: Physiotherapeutic intervention — Participants received one session per week, until a total of 20 sessions were completed: Group 1 (n=20) received the muscle compression treatment. Group 2 (n=20) received the manual massage treatment. Group 3 (n=20) received the hydrotherapy treatment and group 4 (n=20) received the active recovery treatment.
Other: Data Analysis — The usual descriptive parameters (mean and standard deviation) of the sample were calculated. The distribution and analysis of the other data were performed by means of a nonparametric test (Mann-Whitney U test) comparing the groups. A confidence level of 95% was established, considering a value of p<0.05 as statistically significant.

SUMMARY:
Acute fatigue is the inability to generate a required or expected level of force or exercise intensity, whether or not preceded by previous exercise. It is an important risk factor in overuse injuries. It is multifactorial in nature and its mechanisms of formation are imprecise. This type of fatigue can affect both the peripheral level, generating neuromuscular or peripheral fatigue, and the central level, generating central fatigue Objective: To study several physiotherapeutic protocols, analyzing the degree of effectiveness of each one for the recovery of acute fatigue in athletes. Design: Prospective randomized experimental study with 4 groups of physiotherapeutic protocols suitable in acute fatigue recovery. Participants: Presentation of 80 patients treated with 4 therapeutic protocols, equally divided and purposely sexed. The four protocols were divided into: Active recovery (n=20) hydrotherapy (n=20) massage (n=20) and compression (n=20) for 4 weeks of treatment. Intervention: Active recovery protocols (group 1) hydrotherapy protocol (group 2) massage protocol (group 3) and comprehension protocol (group 4).

Keywords: Lower limbs, physiotherapy, athlete, biomechanics, protocol.

DETAILED DESCRIPTION:
The etiology of injury in sport is multifactorial, generated by both intrinsic and extrinsic factors. There is evidence that supports that the management and handling of loads is the factor that generates the greatest risk of injury and that not respecting the load-recovery balance can lead to an accumulation of fatigue resulting in poor training adaptation which leads to increased risk of injury. From a physiological approach, fatigue is defined as a functional failure of the organism which, due to excessive energy expenditure and depletion of substrates necessary for energy production, leads to a decrease in performance.

Acute fatigue is the inability to generate a required or expected level of exercise force or intensity, whether or not preceded by previous exercise. Acute fatigue is an important risk factor in overuse injuries. It is multifactorial in nature and its mechanisms of formation are imprecise. This type of fatigue can affect both the peripheral level, generating neuromuscular or peripheral fatigue, and the central level, generating central fatigue. Peripheral or neuromuscular fatigue is the result of altered musculoskeletal homeostasis due to a limitation or failure of one or more motor unit processes, producing a dysfunction in the contraction process. Central fatigue is an involuntary failure in brain function or nerve impulse conduction, resulting in impaired transmission from the central nervous system (CNS) and impaired motor axon recruitment. One of the main factors associated with central fatigue is the alteration of synthesis and activity of some neurotransmitters.

Elite athletes push their training to the limit in order to maximize their performance. This generates muscle damage that results in a breakdown of structural proteins of muscle fibers and connective tissues, causing tissue inflammation, Delayed Onset Muscle Soreness (DOMS) and an increase in perceived fatigue. To maximize an athlete's ability to perform, it is not only the training that must be addressed, but also the balance between training and recovery. This prevents maladaptation to physiological and psychological stresses induced by the load. Therefore, it is important for the athlete to optimize the recovery period to reduce the risk of injury.

The purpose of this research is to demonstrate the efficacy of various physiotherapeutic protocols, analyzing the degree of effectiveness in each of these for recovery from acute fatigue in athletes.

ELIGIBILITY:
Inclusion Criteria:

* Active athletes
* Presentation of typical clinical signs of acute fatigue in one of the two lower limbs
* Positive diagnosis of acute fatigue

Exclusion Criteria:

* Not compatible with age range
* Healthy athletes
* Diagnosed injuries other than acute fatigue

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Questionnaire (STAI) | five months
  The range or index of anxiety perceived during the exam and the ability to tolerate anxious moments are evaluated.
Rating of Perceived Exertion (RPE) | five months
  The range or rate of perceived exertion during the scan is evaluated.
Scale Countermovement jump (CMJ) | five months
  The range or index of neuromuscular performance during the scan is evaluated.

SECONDARY OUTCOMES:
Number of participants in each physical therapy application | five months
  Five reviews were carried out corresponding to the five months of treatment. During these five months, the participants received one session per week, until a total of 20 sessions were completed:
  * Group 1 (n=20) received the muscle compression treatment.
  * Group 2 (n=20) received the manual massage treatment.
  * Group 3 (n=20) received the hydrotherapy treatment.
  * Group 4 (n=20) received the active recovery treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gema León Bravo, Physiotherap, Principal Investigator — Gema León Physiotherapy and Rehabilitation Clinic; Rafael Arenas Quiles, Physiotherap, Study Chair — Universidad de Córdoba
Locations (1):
- Gema León Physiotherapy and Rehabilitation Clinic, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No
The request for the data will be studied and considered upon prior and justified request.

REFERENCES:
- [Background] Benjaminse A, Webster KE, Kimp A, Meijer M, Gokeler A. Revised Approach to the Role of Fatigue in Anterior Cruciate Ligament Injury Prevention: A Systematic Review with Meta-Analyses. Sports Med. 2019 Apr;49(4):565-586. doi: 10.1007/s40279-019-01052-6. PMID 30659497
- [Background] Guan Y, Bredin S, Jiang Q, Taunton J, Li Y, Wu N, Wu L, Warburton D. The effect of fatigue on asymmetry between lower limbs in functional performances in elite child taekwondo athletes. J Orthop Surg Res. 2021 Jan 9;16(1):33. doi: 10.1186/s13018-020-02175-7. PMID 33422109
- [Background] Burton I. Autoregulation in Resistance Training for Lower Limb Tendinopathy: A Potential Method for Addressing Individual Factors, Intervention Issues, and Inadequate Outcomes. Front Physiol. 2021 Aug 5;12:704306. doi: 10.3389/fphys.2021.704306. eCollection 2021. PMID 34421641
- [Background] Trojian T, Driban J, Nuti R, Distefano L, Root H, Nistler C, LaBella C. Osteoarthritis action alliance consensus opinion - best practice features of anterior cruciate ligament and lower limb injury prevention programs. World J Orthop. 2017 Sep 18;8(9):726-734. doi: 10.5312/wjo.v8.i9.726. eCollection 2017 Sep 18. PMID 28979857
- [Background] Franke TPC, Backx FJG, Huisstede BMA. Lower extremity compression garments use by athletes: why, how often, and perceived benefit. BMC Sports Sci Med Rehabil. 2021 Mar 24;13(1):31. doi: 10.1186/s13102-020-00230-8. PMID 33761989
- [Background] Ghram A, Young JD, Soori R, Behm DG. Unilateral Knee and Ankle Joint Fatigue Induce Similar Impairment to Bipedal Balance in Judo Athletes. J Hum Kinet. 2019 Mar 27;66:7-18. doi: 10.2478/hukin-2018-0063. eCollection 2019 Mar. PMID 30988836
- [Background] Cejudo A, Sainz de Baranda P, Ayala F, De Ste Croix M, Santonja-Medina F. Assessment of the Range of Movement of the Lower Limb in Sport: Advantages of the ROM-SPORT I Battery. Int J Environ Res Public Health. 2020 Oct 19;17(20):7606. doi: 10.3390/ijerph17207606. PMID 33086605
- [Background] DeLang MD, Salamh PA, Farooq A, Tabben M, Whiteley R, van Dyk N, Chamari K. The dominant leg is more likely to get injured in soccer players: systematic review and meta-analysis. Biol Sport. 2021 Sep;38(3):397-435. doi: 10.5114/biolsport.2021.100265. Epub 2020 Oct 28. PMID 34475623
- [Background] Gilbert FC, Burdette GT, Joyner AB, Llewellyn TA, Buckley TA. Association Between Concussion and Lower Extremity Injuries in Collegiate Athletes. Sports Health. 2016 Nov/Dec;8(6):561-567. doi: 10.1177/1941738116666509. Epub 2016 Sep 20. PMID 27587598
- [Background] Drury B, Ratel S, Clark CCT, Fernandes JFT, Moran J, Behm DG. Eccentric Resistance Training in Youth: Perspectives for Long-Term Athletic Development. J Funct Morphol Kinesiol. 2019 Nov 28;4(4):70. doi: 10.3390/jfmk4040070. PMID 33467385
- [Background] Mang CS, Whitten TA, Cosh MS, Dukelow SP, Benson BW. Assessment of Postural Stability During an Upper Extremity Rapid, Bimanual Motor Task After Sport-Related Concussion. J Athl Train. 2020 Nov 1;55(11):1160-1173. doi: 10.4085/1062-6050-378-19. PMID 33064821
- [Background] Avedesian JM, Covassin T, Dufek JS. The Influence of Sport-Related Concussion on Lower Extremity Injury Risk: A Review of Current Return-to-Play Practices and Clinical Implications. Int J Exerc Sci. 2020 Aug 1;13(3):873-889. doi: 10.70252/WVYL1782. eCollection 2020. PMID 32922630
- [Background] Frutuoso AS, Diefenthaeler F, Vaz MA, Freitas Cde L. LOWER LIMB ASYMMETRIES IN RHYTHMIC GYMNASTICS ATHLETES. Int J Sports Phys Ther. 2016 Feb;11(1):34-43. PMID 26900498
- [Background] Siupsinskas L, Garbenyte-Apolinskiene T, Salatkaite S, Gudas R, Trumpickas V. Association of pre-season musculoskeletal screening and functional testing with sports injuries in elite female basketball players. Sci Rep. 2019 Jun 26;9(1):9286. doi: 10.1038/s41598-019-45773-0. PMID 31243317
- [Background] Dubose DF, Herman DC, Jones DL, Tillman SM, Clugston JR, Pass A, Hernandez JA, Vasilopoulos T, Horodyski M, Chmielewski TL. Lower Extremity Stiffness Changes after Concussion in Collegiate Football Players. Med Sci Sports Exerc. 2017 Jan;49(1):167-172. doi: 10.1249/MSS.0000000000001067. PMID 27501359
- [Background] Beck B, Drysdale L. Risk Factors, Diagnosis and Management of Bone Stress Injuries in Adolescent Athletes: A Narrative Review. Sports (Basel). 2021 Apr 16;9(4):52. doi: 10.3390/sports9040052. PMID 33923520